CLINICAL TRIAL: NCT06354582
Title: Effect of Intravenous Vitamin C on Intrapartum Maternal Fever After Epidural Labor Analgesia : A Randomized Controlled Trial
Brief Title: Effect of Intravenous Vitamin C on Intrapartum Maternal Fever After Epidural Labor Analgesia
Acronym: EIVCIMFAELA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kunyue Li (Other)
Collaborators: Third Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor-Investigator, Kunyue Li, Principal Investigator, Third Affiliated Hospital of Zhengzhou University
Organization: Third Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-085-01
Record Dates: First submitted 2024-03-26; First posted 2024-04-09 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Obstetric Labor Complications; Fever
Keywords: Intrapartum maternal fever; Epidural analgesia; Inflammation; Vitamin C
MeSH Terms: conditions — Obstetric Labor Complications; Fever; Inflammation | interventions — Ascorbic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parturients are randomly assigned to either vitamin C(1,2,3) or control. The vitamin C group received 1 g, 2g, and 3g of vitamin C intravenously respectively and the control group received normal saline, administered after the induction of epidural labor anesthesia. There will be 100 cases in each group. The infusion speed will be set at 5ml/min.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group C1 (Experimental): The vitamin C1 group will receive 1 g of vitamin C intravenously administered after the induction of epidural labor anesthesia. The infusion speed will be set at 5ml/min.
  Interventions: Drug: Vitamin C Injection
- Group C2 (Experimental): The vitamin C2 group will receive 2 g of vitamin C intravenously administered after the induction of epidural labor anesthesia. The infusion speed will be set at 5ml/min.
  Interventions: Drug: Vitamin C Injection
- Group C3 (Experimental): The vitamin C3 group will receive 3 g of vitamin C intravenously administered after the induction of epidural labor anesthesia. The infusion speed will be set at 5ml/min.
  Interventions: Drug: Vitamin C Injection
- Group P (Placebo Comparator): The control group P will receive normal saline and be administered after the induction of epidural labor anesthesia. The infusion speed will be set at 5ml/min.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Vitamin C Injection — Drug Specification: 5ml: 1g. Method: parturients in each group will be intravenously injected with corresponding dose after receiving epidural labor analgesia.
  Other Names: Suicheng, H20046552
  Arms: Group C1; Group C2; Group C3
Other: Normal saline — The placebo comparator will receive normal saline with the same volume and be administered after the induction of epidural labor anesthesia.
  Arms: Group P

SUMMARY:
This study aims to explore the effect of intravenous vitamin C infusion on intrapartum fever after epidural labor analgesia, to reduce the impact of intrapartum fever on maternal and infant, improve maternal and infant outcomes, and provide a reference for clinical preventive medication.

DETAILED DESCRIPTION:
Parturients who request pain relief would receive epidural labor analgesia after the obstetrician and anesthesiologist jointly evaluated and approved. The epidural catheter was inserted at the intervertebral space of either L2-3 or L3-4. 5 ml 1.5% chloroprocaine (with 1:200,000 epinephrine) as a test was delivered to parturients via the catheter. Then parturients would be observed for 5 min whether there were adverse reactions and then were given an initial dose of 10 ml ropivacaine 0.08% with sufentanil 0.3 µg/ml. After that, a patient-controlled epidural analgesia (PCEA) pump (240ml 0.08% ropivacaine with sufentanil 0.3 µg/ml) would be attached to the catheter. The pump would be set to administer an 8 ml bolus every 20 minutes and a 2 ml patient-controlled bolus with the same interval. Subsequently, trained nursing staff would take charge of the parturients and inform the obstetrician. The basic condition of parturients was monitored during the whole process. After that, parturients in each group will be administered vitamin C intravenously except the group for placebo-controlled.

ELIGIBILITY:
Inclusion Criteria:

* single-fetus, head position, and full-term vaginal delivery receiving epidural labor analgesia.

Exclusion Criteria:

* have a fever before epidural analgesia, acute infection on admission, incomplete baseline data, fatal fetal malformations or comorbidities, duration from admission to delivery of more than 72 hours or less than 3 hours, or an American Society of Anesthesiologists (ASA) classification of ≥ Ⅲ.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Intrapartum fever or not | Every two hours after receiving epidural labor analgesia, until baby delivery
  The temperature of parturients ≥ 37.5℃
The temperature of parturients | Every two hours after receiving epidural labor analgesia, until baby delivery.
  After receiving epidural labor analgesia
The duration of intrapartum fever | Every two hours after receiving epidural labor analgesia, until baby delivery.
  If parturients develop intrapartum fever, record the lasting time of fever.
Complete blood count indicators | Take blood test immediately before analgesia, immediately when parturients is developing intrapartum fever and immediately after delivery
  Record the blood cell indicators for three times totally

SECONDARY OUTCOMES:
Visual analogue scale(VAS) | Every two hours after receiving epidural labor analgesia, until baby delivery.
  Record the Visual analogue scale(VAS) of parturients at every time point. The visual analogue scale scores ranged from 0 to 10, with higher scores indicating increased pain levels.
Amount of total analgesics | immediately After the baby is delivered
  Record the amount of total analgesics
Side effects on mothers | immediately After the baby is delivered
  Record the incidence of pruritus, vertigo, prosthesis, dyspnea, nausea and vomiting of parturients
the duration of total labor | immediately After the baby is delivered
  Delivery characteristics 1
Incidence of rupture of membranes | immediately After the baby is delivered
  Delivery characteristics 1
Delivery characteristics 2 | immediately After the baby is delivered
  Record the incidence of lateral vaginal incision, postpartum hemorrhage, amniotic fluid contamination.
Record the weight of the baby. | immediately After the baby is delivered
  Infant characteristics 1
Record the gender of the baby. | immediately After the baby is delivered
  Infant characteristics 2
Apgar score | immediately After the baby is delivered
  Record the 1min, 5min Apgar score of the baby.
the incidence of fetal distress | immediately After the baby is delivered
  Infant characteristics 4
Record the infant ward administration. | immediately After the baby is delivered
  Infant characteristics 4

CONTACTS AND LOCATIONS:
Overall Officials: Tao Wang, PhD, Study Director — the Third Affilated Hospital of Zhengzhou University
Locations (1):
- Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
We will upload our main outcomes, study protocol, and statistical methods on this platform after all the work is done, and further inquiries can be directed to our investigators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start from January, 2026 to April, 2026.
Access Criteria: At this platform and further send e-mail to investigators.

REFERENCES:
- [Result] Patel S, Ciechanowicz S, Blumenfeld YJ, Sultan P. Epidural-related maternal fever: incidence, pathophysiology, outcomes, and management. Am J Obstet Gynecol. 2023 May;228(5S):S1283-S1304.e1. doi: 10.1016/j.ajog.2022.06.026. Epub 2023 Mar 14. PMID 36925412
- [Result] Sultan P, Segal S. Epidural-Related Maternal Fever: Still a Hot Topic, But What Are the Burning Issues? Anesth Analg. 2020 Feb;130(2):318-320. doi: 10.1213/ANE.0000000000004576. No abstract available. PMID 31934906
- [Result] Hensel D, Zhang F, Carter EB, Frolova AI, Odibo AO, Kelly JC, Cahill AG, Raghuraman N. Severity of intrapartum fever and neonatal outcomes. Am J Obstet Gynecol. 2022 Sep;227(3):513.e1-513.e8. doi: 10.1016/j.ajog.2022.05.031. Epub 2022 May 19. PMID 35598690
- [Result] Morton S, Kua J, Mullington CJ. Epidural analgesia, intrapartum hyperthermia, and neonatal brain injury: a systematic review and meta-analysis. Br J Anaesth. 2021 Feb;126(2):500-515. doi: 10.1016/j.bja.2020.09.046. Epub 2020 Nov 18. PMID 33218673